CLINICAL TRIAL: NCT03347227
Title: Characterization of Arrhythmia Substrate to Ablate Persistent Atrial Fibrillation (Coast-AF) Randomized Clinical Trial
Brief Title: Characterization of Arrhythmia Substrate to Ablate Persistent Atrial Fibrillation
Acronym: COAST-AF RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: AF ablation; Pulmonary vein isolation; Atrial scar ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Prospective, parallel arm randomized clinical trial
Who Masked: Participant
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Vein Isolation (Active Comparator): Wide area circumferential catheter ablation for pulmonary vein isolation
  Interventions: Procedure: Catheter ablation
- Pulmonary Vein Isolation and scar ablation (Experimental): Wide area circumferential catheter ablation for pulmonary vein isolation and scar ablation
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — Wide area circumferential catheter ablation for pulmonary vein isolation of persistent atrial fibrillation
  Other Names: Atrial Fibrillation Ablation

SUMMARY:
A multicentre, parallel group, two arm, single-blinded randomized clinical trial, assessing the efficacy of a patient-tailored catheter ablation (CA) strategy guided by atrial scar mapping in addition to pulmonary vein isolation (PVI) when compared to PVI alone in patients with persistent atrial fibrillation (AF).

DETAILED DESCRIPTION:
The optimal CA strategy for persistent AF remains unknown. Current data highlight the need for a better understanding of the substrate and mechanisms of arrhythmia maintenance in this population. Atrial scar-based catheter ablation has recently emerged as a promising strategy for ablation of AF. However, the available data has limitations that preclude definitive conclusions regarding the utility of this strategy (no data from multicenter, randomized studies available). Further research is needed to assess the role of scar-based ablation for persistent AF.

The Investigators hypothesize that catheter ablation of persistent AF (PeAF) tailored to abolish abnormal atrial substrate identified by intracardiac atrial scar mapping in addition to pulmonary vein isolation (PVI) will result in higher procedural success rates when compared to PVI alone.

The study will recruit 502 patients with PeAF (251 per treatment arm) who are candidates for CA ablation of AF according to the treating physician (and in agreement with current practice guidelines). Subjects will be recruited over a 42 month period. The total duration of the study is 60 months.

Prior to undergoing catheter ablation subjects will be seen by the investigator/ research assistant and the following data will be collected:

i. Age and sex ii. Structural heart disease if present iii. CHADS2VASc score iv. DR-FLASH score v. NYHA class vi. Current medications vii. Duration of uninterrupted AF viii. Height and weight ix. Echocardiogram and other cardiac imaging results (within previous 12 months, including assessment of left ventricular ejection fraction, left atrial volume and valve function) x. ECG, Holter or loop monitor recording (within past 36 months) documenting AF.

Subjects will be randomly assigned in a 1:1 ratio to undergo wide area circumferential ablation for pulmonary vein isolation (PVI- control arm) or wide area circumferential ablation PVI and scar ablation (experimental arm). Randomization will be stratified by centre and by sex. Subjects will be randomized prior to the procedure.

Enrolled subjects will have a clinical follow-up visit at 3, 6, 12 and 18 months after the ablation procedure. A 14-day continuous ambulatory ECG monitor will be completed at each visit. The results of monitoring will be interpreted at a centralized core lab, and the results will be adjudicated by an arrhythmia specialist blinded to treatment group. A total of three questionnaires will be administered throughout the study, each at a specific time point. The Quality of Life (EQ-5D), CCS-Severity of AF scale, and Atrial Fibrillation Effect on Quality of life (AFEQT) will be completed at baseline, and at the 12-month and 18 month visit.

Concomitant medical therapy will be selected according to the treating physician. All subjects will be maintained on systemic oral anticoagulation for at least 2 months following catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years ;
2. Subjects with symptomatic persistent AF AND clinically indicated catheter ablation for AF
3. At least one episode of AF that is sustained beyond 3 months in duration ; documented on 12-lead ECG, Holter monitor, loop monitor or trans-telephonic monitor (TTM) within 36 months of enrollment in the study;
4. Modified DR-FLASH score >=4

4. Subjects must be able to provide informed consent.

Exclusion Criteria:

1. History of previous catheter ablation for AF or left atrial flutter;
2. History of previous surgical ablation for AF;
3. Known intracardiac thrombus;
4. Contraindication to systemic oral anticoagulation therapy;
5. Reversible causes of AF;
6. Hypertrophic cardiomyopathy;
7. Severe valvular disease (mitral/aortic stenosis or regurgitation);
8. Subjects that are pregnant or breastfeeding;
9. Comorbid condition with life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2018-08-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of documented (>30s) AF, atrial flutter or atrial tachycardia occuring from day 91 to 18 months post ablation | day 91 post ablation to 18 months
  Documented AF, Aflutter or AT by ECG, holter or external loop monitoring and has a duration of at least 30 seconds

SECONDARY OUTCOMES:
AF burden | At 12 months and 18 months
  Documented amount of AF
Need for repeat ablation procedure for AF, AFl or AT | Up to 18 months
  Documented by ECG, holter or ECG loop recorder
Need for emergency room visits or hospitalization | Up to 18 months
  Hospital admission for > 24 hours and emergency room admission
Incidence of any ECG documented AF with 90 days of ablation | up to 90 days
  Symptomatic or asymptomatic AF
Time to first recurrence at 18 months according to sex and atrial scar extent | 18 months
  Recurrence of AF, AFl or AT
Composite safety outcome | Up to 18 months
  Procedure related complications at any time (stroke, PV stenosis, pericarditis, cardiac perforation, major bleeding) and/or death
Total ablation delivery time | Day of ablation procedure
  RF ablation time
Total procedure duration | Day of ablation procedure
  Start of ablation to end of ablation
Quality of life analyses | 18 months
  Using EQ-5D general quality of life score, and AF severity scale (symptoms and functionality)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Nery, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (15):
- Canada (15):
  - Libin Cardiovascular Institute, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - QEII Health Sciences Centre, Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Rouge Valley Regional Heart Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Sacre-Coeur Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Institute Universitaire de Cardiologie et Pneumologie du Quebec (IUCPQ), Québec, Quebec
  - CIUSSS de L'Estrie-CHUS-Hopital Fleurimont, Sherbrooke, Quebec